CLINICAL TRIAL: NCT06098443
Title: Acupressure Versus Transcutaneous Electrical Nerve Stimulation on Pain and Quality of Life Intradialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed El-Moatasem Mohamed, lecturer of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004482
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2023-12

CONDITIONS: Hemodialysis Complication
MeSH Terms: interventions — Acupressure; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Acupressure (Experimental): The acupressure points will be determined, patients are informed that they will feel soft vibrations and pain during acupressure application. Patients are advised that it is sufficient for them to feel the vibrations of the acupressure device slightly. It be felt first symmetrically right knee, right leg, left knee, left leg Patients will receive acupressure 24 sessions three times a week for eight weeks. After application the patient will be asked about the severity of pain half an hour after administration (Çevik & Taşcı, 2020).
  Interventions: Other: Acupressure
- Transcutaneous electrical nerve stimulation (Active Comparator): • Placement electrodes applied on the painful area lower leg.
  Settings:
  * Intensity up to patient tolerance.
  * Duration 30min.
  Interventions: Device: Transcutaneous electrical nerve stimulation

INTERVENTIONS:
Other: Acupressure — Acupressure is effective on anxiety and depression management. acupressure therapy at K1, ST36, and SP6 acupoints significantly reduced anxiety & depression in patients with ESRD.
  Arms: Acupressure
Device: Transcutaneous electrical nerve stimulation — TENS lead to meaningful reduction of pain in patients suffering from difficult to treat phantom limb pain. This treatment has a high success rate and is associated with high satisfaction rates and no reported adverse events. The suggested duration of treatment is at least 30 minutes and may be extended up to 45 minutes. TENS delivers pulsed electric currents across the intact surface of the skin to stimulate peripheral nerves and the spinal cord, resulting in segmental and extra segmental analgesia. TENS delivers pulsed electric currents across the intact surface of the skin to stimulate peripheral nerves and the spinal cord, resulting in segmental and extrasegmental analgesia. (Vathakul et al., 2022).
  Arms: Transcutaneous electrical nerve stimulation

SUMMARY:
Hemodialysis patients have a high prevalence of pain, mainly musculoskeletal and intra dialytic pain. A high prevalence of pain was also observed in the upper and lower limbs and the trunk. In addition, severe functional interference of pain in the ability to walk was associated with pain in the upper Limb. These results indicate that pain in hemodialysis patients is limiting and disabling (Dos Santos et al., 2021).

Acupressure increases relaxation, relieves pain, and reduces anxiety and depression, especially in the elderly. It is relatively inexpensive, safe, non-invasive, and easy to use and is performed by hands, elbows. by applying pressure to specific areas of the body so muscle spasms are relieved, blood circulation and vital energy are improved (Bastani et al.,2022).

Strong non-painful TENS within or close to the site of pain produces clinically important reductions in the intensity of pain during or immediately after treatment. With no reports of serious adverse events. TENS as an adjunct to core treatment or immediate short-term relief of pain, irrespective of diagnosis. Patients should be advised to tailor TENS Treatment according to their individual needs (Johnson et al., 2022).

DETAILED DESCRIPTION:
Sixty patients will be randomly assigned into two equal groups (n=30):

1. Group A (30 patients) will receive Acupressure three times per week for eight weeks.
2. Group B (30 patients) will receive TENS three times per week for eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* • Sixty patients with renal failure stage 5 undergoing hemodialysis sessions at least six months ago up to 2 years.

  * Participants with lower limb pain and brief pain inventory (BPI) pain score between 7 and 10 points.
  * Body mass index ranges from 25 to 29.9.
  * Their ages range from 50-60 years old.
  * All patients will be under full medical control.
  * Patients will be free from lower limb dialysis grafting.
  * Hemoglobin level more than 10 mg\dl.

Exclusion Criteria:

* Skin disease such as dermatitis, stitches and wound.
* Active infection, autoimmune diseases and malignancy.
* Severe cardiac diseases.
* Severe chest diseases.
* Patients with cardiac pacemaker.
* Epilepsy.
* Using another integrative treatment method during the study.
* Uncontrolled diabetes.
* Deep vein thrombosis.
* Lumber disc prolapses affect lower limb.

Ages: 50 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Pain pressure algometry: | Pain pressure algometry:will be measured at baseline, and it will be measured again after eight weeks
  Pain pressure algometry: Device to measure the intensity of painful stimuli objectively
The Brief Pain Inventory (BPI): | The Brief Pain Inventory (BPI): will be measured at baseline, and it will be measured again after eight weeks
  The Brief Pain Inventory (BPI): Is a multidimensional pain assessment tool used to evaluate pain severity and pain interference. The BPI has been translated and validity estimated across multiple languages and patient populations for clinical and research settings.
Short form -36 questionnaire (KDQoL SF-36): | Short form -36 questionnaire (KDQoL SF-36):will be measured at baseline, and it will be measured again after eight weeks
  Short form -36 questionnaire (KDQoL SF-36): Is generic measure of health that has also been used widely in trials in hemodialysis patients for the objective measure quality of life

SECONDARY OUTCOMES:
The incremental shuttle walking test (ISWT): | The incremental shuttle walking test (ISWT):will be measured at baseline, and it will be measured again after eight weeks
  The incremental shuttle walking test (ISWT):Is an important marker of aerobic capacity in patients on renal dialysis
Patient health questionnaire PHQ-9: | Patient health questionnaire PHQ-9:will be measured at baseline, and it will be measured again after eight weeks
  Patient health questionnaire PHQ-9: Is a nine-item questionnaire designed to screen depression in primary care and other medical settings

CONTACTS AND LOCATIONS:
Overall Officials: Hany Obaya, assistant professor, Principal Investigator — giza, Egypt, 12511
Locations (1):
- Cairo University, Cairo, Egypt